CLINICAL TRIAL: NCT07045818
Title: DLPFC Desynchronization and Sympathetic Cardiac Hyperarousal During Aversive Emotional Processing in Women With Recurrent Pregnancy Loss and Comorbid Anxiety: a Multimodal fNIRS-ECG Study (NEURO-CARD-fNIRS)
Brief Title: DLPFC and Sympathetic Reactivity in RPL With Anxiety
Status: Recruiting | Type: Observational
Sponsor: Shenyang Medical College (Other)
Collaborators: Central Hospital Affiliated to Shenyang Medical Collage (Other); The Second Hospital of Shenyang Medical College (Other)
Responsible Party: Principal Investigator, Lin Tao, Assoc. Prof., Shenyang Medical College
Other Study IDs: NEURO-CARD-fNIRS
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Pregnancy Loss Without Current Pregnancy; Anxiety Disorder
Keywords: recurrent pregnancy loss; anxiety; emotion-autonomic dysregulation; dorsolateral prefrontal cortex; functional near-infrared spectroscopy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with recurrent pregnancy loss and comorbid anxiety: Following comprehensive obstetric and psychiatric assessment, participants will be assigned to the "recurrent pregnancy (RPL) with anxiety" or "RPL without anxiety" group based on DSM-5 diagnosis of at least one core anxiety disorder (generalized anxiety disorder, panic disorder, social anxiety disorder, or post-traumatic stress disorder).
  Interventions: Behavioral: Emotional provocation task involving multisensory aversive stimuli
- Women with recurrent pregnancy loss without comorbid anxiety: Following comprehensive obstetric and psychiatric assessment, participants will be assigned to the "RPL with anxiety" or "RPL without anxiety" group based on DSM-5 diagnosis of at least one core anxiety disorder (generalized anxiety disorder, panic disorder, social anxiety disorder, or post-traumatic stress disorder).
  Interventions: Behavioral: Emotional provocation task involving multisensory aversive stimuli

INTERVENTIONS:
Behavioral: Emotional provocation task involving multisensory aversive stimuli — To elicit hemodynamic responses in the dorsolateral prefrontal cortex (DLPFC) and activate the sympathetic nervous system, we used a standardized multisensory aversive stimulation protocol comprising: (i) Visual stimuli: 72 high-arousal images from the GAPED database (moral violations, legal violations, fear-related) shown in 12 blocks (6 images/block, 5 s each) with 20 s baseline and 30 s stimulation; (ii) Auditory stimuli: each block paired with 30 s of calibrated 90 dB(A) high-frequency narrowband white noise (4 kHz center frequency), shown to increase heart rate; (iii) Cold-pain stimuli: during each block, participants placed both hands on 0 °C ice-filled bottles for pain-induced sympathetic activation. This tri-modal task reliably provokes DLPFC engagement and autonomic responses.

SUMMARY:
We propose an exploratory clinical study (NEURO-CARD-2) that employs simultaneous functional near-infrared spectroscopy (fNIRS) and electrocardiography (ECG) to investigate interhemispheric dysfunction in the dorsolateral prefrontal cortex (DLPFC) and its relationship with autonomic sympathetic activation in women with recurrent pregnancy loss (RPL) and comorbid anxiety. Using a standardized multisensory aversive emotional stimulation paradigm, the study will assess cortical and cardiac responses within the framework of the Brain-Heart-Emotion interaction model. The objective is to identify neurobiological signatures underlying emotion-autonomic dysregulation in this population, thereby informing future development of precision-targeted interventions.

DETAILED DESCRIPTION:
Recurrent pregnancy loss (RPL), defined as two or more consecutive pregnancy losses before 24 weeks' gestation, affects an estimated 2-5% of reproductive-aged couples worldwide. Beyond its profound reproductive consequences, RPL carries a heavy psychological burden: approximately 50% of affected women experience chronic anxiety. This emotional distress is more than a mental health concern-it triggers persistent sympathetic activation, evidenced by elevated resting heart rate and diminished heart rate variability (HRV), thus compounding cardiovascular and reproductive risks in a self-reinforcing pathogenic cycle.

Modern psycho-cardiology paradigms, backed by statements from the American Heart Association, underscore the intimate interplay between emotional dysregulation and autonomic dysfunction. Yet the neural mechanisms linking altered central emotion regulation to cardiac autonomic outcomes in women with RPL remain largely elusive-especially in those with comorbid anxiety.

Emerging theories in interoceptive neuroscience suggest that higher-order brain regions could serve as shared neural substrates mediating both anxiety and sympathetic overactivation. In particular, the dorsolateral prefrontal cortex (DLPFC), a critical node within the cognitive control and central autonomic networks, stands out. Evidence from neuroimaging and neuromodulation studies demonstrates hemispheric asymmetry in the DLPFC: the right DLPFC is implicated in threat processing, anxiety generation, and sympathetic arousal, whereas the left DLPFC supports cognitive reappraisal, emotional inhibition, and parasympathetic modulation.

We propose a Brain-Heart-Emotion interaction model in which effective and adaptive autonomic responses depend on synchronized bilateral activation of the DLPFC during negative emotional challenge. Conversely, functional decoupling-manifested as right-lateralized DLPFC dominance-may undermine emotion regulation capacity and precipitate sympathetic overdrive. In women with RPL and comorbid anxiety, this decoupling is posited to drive the convergence of emotional dysregulation and cardiac dysfunction, thereby elevating the risk of adverse reproductive and cardiovascular outcomes.

To test this hypothesis, we have designed a prospective, exploratory clinical study employing simultaneous functional near-infrared spectroscopy (fNIRS) and electrocardiography (ECG) during a standardized multisensory emotional provocation paradigm. We will investigate patterns of interhemispheric DLPFC activation and their relationship to heart rate dynamics in women with recurrent pregnancy loss (RPL), in the presence versus absence of comorbid anxiety, within the proposed Brain-Heart-Emotion framework.

If confirmed, these findings will provide both mechanistic insight and empirical justification for neurobiologically informed, precision-targeted interventions. In particular, they may support the application of inhibitory neuromodulation targeting the right DLPFC, with the potential to deliver multidimensional therapeutic benefits-including enhanced emotional regulation, restoration of autonomic balance, reduced long-term cardiovascular risk, and improved reproductive outcomes in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-45 years, right-handed;
* Diagnosis of recurrent pregnancy loss-defined as ≥2 consecutive spontaneous miscarriages before 28 weeks' gestation;
* Not currently pregnant, or diagnosed with missed abortion at the time of assessment;
* Completed structured psychiatric evaluation by licensed psychiatrists at each center, with diagnostic confirmation per DSM-5.

Exclusion Criteria:

* Use of psychotropic medications in the past month (e.g., SSRIs, SNRIs, TCAs, benzodiazepines, antipsychotics, mood stabilizers);
* Unstable or uncontrolled hypertension (SBP > 180 mmHg or < 90 mmHg);
* Major comorbid organic conditions (e.g., hyperthyroidism, atrial fibrillation, valvular heart disease, stroke, epilepsy, traumatic brain injury, chronic pulmonary disease);
* Significant sensory or communication barriers (e.g., hearing impairment, language difficulty, sensory neuropathy) that could impair task performance or stimulus perception;
* High suicide risk or severe psychiatric comorbidity (e.g., schizophrenia, bipolar disorder, psychotic disorders, substance use disorders);
* Extreme intolerance to auditory, visual, or cold stimuli, based on medical history or pre-test report;
* Any other condition judged by the research physician to interfere with participation in the multisensory emotional stimulation protocol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with recurrent pregnancy loss
Study Population: Recruitment is expected to occur through obstetrics and gynecology outpatient clinics, as well as community outreach via flyers and media campaigns.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Interhemispheric asymmetry of DLPFC activation during aversive emotional stimulation (group × hemisphere interaction). | Single-session fNIRS-ECG protocol
  The primary outcome is the interaction between diagnostic group (RPL with anxiety vs RPL without anxiety) and hemisphere (right vs left dorsolateral prefrontal cortex, DLPFC) in response to aversive emotional stimulation, assessed using a linear mixed-effects model (LME). The model includes fixed effects for group, hemisphere, and their interaction, with random intercepts specified for participants. Post hoc pairwise comparisons of estimated marginal means are conducted using linear contrasts, and Bonferroni correction is applied to account for multiple comparisons. We hypothesise that participants with RPL and comorbid anxiety will exhibit significantly greater right-lateralised DLPFC activation relative to those without anxiety, reflecting altered interhemispheric asymmetry in emotion regulation pathways.

SECONDARY OUTCOMES:
Group difference in interhemispheric synchronization of DLPFC activity | Single-session fNIRS-ECG protocol
  Interhemispheric synchronization in the dorsolateral prefrontal cortex (DLPFC) is assessed using wavelet transform coherence (WTC) between homologous fNIRS channels. Coherence values are averaged across the frequency band of interest (0.01-0.08 Hz) and time window, background-corrected using the 3-minute resting period, and Fisher z-transformed. Group-level statistical comparisons will be then performed on the resulting z-values.
Group difference in averaged heart rate increase during aversive emotional stimulation | Single-session fNIRS-ECG protocol
  For time-domain heart rate variability analysis, preprocessed R-R intervals are resampled at 11 Hz and filtered using a 4th-order low-pass Butterworth filter (cutoff: 0.1 Hz) to suppress respiratory and cardiac noise. Data will be segmented into 40-second epochs (10 s pre-stimulation and 30 s stimulation), and baseline correction will be applied. Mean heart rate elevation during stimulation is computed for each of the 12 blocks and averaged per participant. Between-group comparisons will be performed on the resulting values.

OTHER OUTCOMES:
Joint clustering of interhemispheric wavelet transform coherence (WTC) values and heart rate response features | Single-session fNIRS-ECG protocol
  Unsupervised K-means clustering (k = 2) will be performed on a combined feature space comprising interhemispheric wavelet transform coherence (WTC) values from DLPFC HbO signals and heart rate change metrics. This approach aims to reveal distinct neurobiological phenotypes that differentiate RPL women with comorbid anxiety from those without.
  The resulting cluster structure will be depicted using 95 % confidence ellipses, with cluster centroids indicated by an "X." Alignment between data-driven clusters and predefined clinical groups ("RPL with anxiety" vs "RPL without anxiety") will be quantified using the Adjusted Rand Index (ARI). Finally, cluster separability in this two-dimensional space will be statistically evaluated via Hotelling's T² test.
Comparison of adverse events (AEs) and serious adverse events (SAEs) between groups | Single-session fNIRS-ECG protocol
  AEs include any signs of discomfort, distress, or autonomic instability during stimulation (e.g., acute anxiety, withdrawal requests). SAEs are defined as events such as syncope, extreme anxiety episodes, or severe physiological reactions requiring clinical intervention. All adverse events will be monitored in real time by trained researchers and documented per predefined criteria. Group-level differences in AE and SAE incidence will be descriptively analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-En Liu, MD, Study Chair — Shenyang Medical College; Lin Tao, MM, Principal Investigator — Shenyang Medical College; Fei Meng, MD, Study Director — Central Hospital Affiliated to Shenyang Medical Collage; Xiu-Ling Zhang, MD, Study Director — The Second Hospital of Shenyang Medical College
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Shenyang Medical College, Shenyang, Liaoning
  - Central Hospital Affiliated to Shenyang Medical Collage, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: Yes
De-dentified individual participant data, together with the full study protocol, MATLAB analysis scripts, and all supporting materials, will be released in full at the time of publication of the final manuscript. All materials will be deposited on one internationally recognized open science repository selected by the research team, such as Open Science Framework (https://osf.io), Zenodo (https://zenodo.org), or GitHub (https://github.com). Access will be granted for non-commercial research purposes. Requests for additional information may be directed to the corresponding author.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Available at the time of publication of the final article
Access Criteria: Data will be deposited on the Open Science Framework (https://osf.io) and will be accessible for non-commercial research purposes.